CLINICAL TRIAL: NCT07091955
Title: Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy of a Probiotic Preparation in the Prevention of Upper Respiratory Tract Infections in a Healthy Adult Population
Brief Title: Clinical Trial to Evaluate the Efficacy of a Probiotic Preparation in the Prevention of Upper Respiratory Tract Infections in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioithas SL (Industry)
Collaborators: Centro Sperimentale del Latte S.r.l. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRESP.PROB
Record Dates: First submitted 2025-07-08; First posted 2025-07-29 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: URTI - Viral Upper Respiratory Tract Infection; Prevention
Keywords: upper respiratory tract infections; prevention; probiotics; microbiota; microbiome
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled with parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lacticaseibacillus rhamnosus CRL1505 (Experimental): Probiotic product containing Lacticaseibacillus rhamnosus CRL1505 formulated in a vegetable hydroxymethylpropyl-cellulose capsule of size 2
  Interventions: Dietary Supplement: Lacticaseibacillus rhamnosus CRL1505
- Placebo (Placebo Comparator): Placebo product containing cornstarch, in a vegetable hydroxymethylpropyl-cellulose capsule of size 2
  Interventions: Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Lacticaseibacillus rhamnosus CRL1505 — Probiotic product containing Lacticaseibacillus rhamnosus CRL1505 formulated in a vegetable hydroxymethylpropyl-cellulose capsule of size 2
  Arms: Lacticaseibacillus rhamnosus CRL1505
Dietary Supplement: Placebo Comparator — Placebo product containing cornstarch, in a vegetable hydroxymethylpropyl-cellulose capsule of size 2
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo-controlled, parallel-group, clinical trial to assess the efficacy of the intake of a probiotic product composed of Lacticaseibacillus rhamnosus CRL1505 strain in reducing or preventing upper respiratory tract infections (URTIs) in a healthy adult population

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, parallel-group, clinical trial. The study aims to demonstrate the efficacy of the intake of a probiotic product composed of Lacticaseibacillus rhamnosus CRL1505 strain in reducing or preventing upper respiratory tract infections in a healthy adult population.

The study will be focused on a healthy population, so the exclusion criteria will rule out individuals with major acute or chronic illnesses and an immunocompromised state. In addition, those subjects with a regular pharmacological treatment or consumption of food supplements that could influence the outcome of the study in the last 4 weeks prior to inclusión will be excluded. If patients could discontinue this treatment after a washout period and during the intervention period, they would be able to participate in the study. However, the usual medication that is considered not to influence the results of the study will be allowed. Subjects recently vaccinated against influenza will also be excluded, but as the study focuses on a healthy population, a priori vaccination is not recommended and there would be no problem in finding subjects with these characteristics because there is no contradiction.

In addition, subjects included will be asked not to modify their diet or physical activity during the study.

An important data that is not usually recorded in many studies is the use of medication to alleviate the symptoms of URTI, either non-prescription or prescribed by the physician. Only antibiotic medication to treat or prevent bacterial upper respiratory tract coinfections or complications is usually established as a variable (the use of antibiotics is established as a secondary variable in the present study). The investigators consider that it is very important to record the use of these treatments to evaluate if any study group is unbalanced in this regard and/or whether it is a confusion factor when interpreting the results. The investigators could consider the possibility of performing a post hoc analysis of this topic and present it in the final report if the results are interesting.

Similarly, it is important to collect baseline data related to the type of work or continuous contact with people with risk factors such as children or elderly to assess whether the groups are balanced. It will also be collected data about the number of URTIs in the study subjects since 3 months prior to inclusion.

The treatment period will be 12 weeks. There will then be a follow-up period (without treatment) of 4 weeks to evaluate the sustained effect of the probiotic product. The study will be structured in 3 face-to-face visits at week 0, 12 and 16.

For the evaluation of the efficacy variables, a diary would be provided to the study subject for a daily evaluation. Saliva collection kits for the determination of salivary IgA in the initial o final visits will also be provided.

The complete inclusion process will be carried out in October and November so that the study was located in the months of highest URTI incidence.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between 18 and 65 years.
* Signed Informed Consent to participate in the study
* BMI less than 35 kg/m2

Exclusion Criteria:

* Chronic pathological conditions such as chronic respiratory diseases (asthma, chronic bronchitis, chronic obstructive pulmonary disease etc), chronic heart diseases (chronic heart failure etc), chronic neurological diseases (Parkinson´s diseases, multiple esclerosis etc), chronic liver diseases, kidney liver diseases, gastrointestinal diseases, hematologic disorders etc, or other disease or condition that the researcher considers
* Metabolic disorders (diabetes, obesity with BMI greater than 35.1 kg/m2 etc).
* Congenital or acquired immune defects (including allergies).
* Immunocompromised individuals (HIV infection, chemotherapy, post-trasplant, chronic corticosteroid treatment etc).
* Presence of nasal ulcers/nasal polyps or other conditions that could cause nasal obstruction.
* Abuse of alcohol, tobacco or other drugs.
* Pregnancy or lactation.
* Regular intake of products that could influence the study outcome (immune suppressants/immune stimulants including paramedication such as Echinacea, analgesics, antiinflammatories, antitussives/expectorants, influenza remedies, mouth or throat therapeutics, decongestants, antibiotics, antihistaminergic drugs, probiotics) within the last 4 weeks prior to the study start.
* Influenza vaccination in the last 6 monts.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Patients who were diagnosed with at least 1, 2 or 3 URTIs | 16 weeks
  Difference in the proportion of patients who were diagnosed with at least 1, 2 or 3 URTIs during the intervention (12 weeks) and follow-up period (16 weeks) between the study groups
Number of URTIs per patient | 16 weeks
  Difference in the mean number of URTIs per patient between the study groups during the intervention period (12 weeks) and follow-up period (16 weeks)
Patients who were diagnosed of common cold and influenza | 16 weeks
  Difference in the proportion of patients who were diagnosed of common cold and influenza during the intervention (12 weeks) and follow-up period (16 weeks) between the study groups.

SECONDARY OUTCOMES:
Participants who presented URTI complications | 16 weeks
  Difference in the proportion of participants who presented URTI complications such as pneumonia, otitis media and acute sinusitis during intervention and follow-up periods between study groups
Number of URTI complications | 16 weeks
  Difference in the number of URTI complications such as pneumonia, otitis media and acute sinusitis during intervention and follow-up periods between study groups
Number of days until the occurrence of the first URTI episode | 12 weeks
  Mean number of days until the occurrence of the fist URTI episode during the 12 week intervention period
Number of days with URTI episode per participant | 16 weeks
  Difference in the mean number of days with URTI episode per participant (days with URTI/number of participants) during the study (12 weeks treatment period and 16 weeks follow-up period)
Duration of URTI episode | 16 weeks
  Difference in the mean duration of each episode of URTI (days with URTI/number of URTIs) during the study, including the treatment period (12 weeks) and the follo-up (16 weeks)
URTI-Free Time Rate | 16 weeks
  Difference in the URTI-Free Time Rate, defined as the proportion of accumulated days where patients do not experience URTIs in relation to the total days of all study (intervention period of 12 weeks and follo up period of 16 weeks)
Participants who presented gastrointestinal infections | 16 weeks
  Difference in the proportion of participants who presented gastrointestinal infections at the intervention and follow-up periods between study groups
Number of gastrointestinal infections | 16 weeks
  Difference in the number of gastrointestinal infections at the intervention and follow-up periods between study groups
Salivary IgA concentrations | 12 weeks
  Difference in mean salivary IgA concentrations during intervention period between study groups
Participants using antibiotics | 16 weeks
  Difference in the proportion of participants using antibiotics during intervention and follow-up periods between study groups
Number of days with antibiotics treatment | 16 weeks
  Difference in the days with antibiotics treatment during intervention and follow-up periods between study groups
Participants using symptomatic treatment | 16 weeks
  Difference in the proportion of participants using symptomatic treatment during intervention and follow-up periods between study groups
Number of days with symptomatic treatment during the study | 16 weeks
  Difference in the days with symptomatic treatment during intervention and follow-up periods between study groups
"Common cold episode day" Wisconsin Upper Respiratory Symptom Survey - 21 item score (WURSS-21 score) | 16 weeks
  Difference in mean "common cold episode day" WURSS-21 score during intervention and follow-up periods between study groups.
  The WURSS-21 score is a validated patient-reported outcome measure designed to assess the impact of upper respiratory tract infections (URTI), such as the common cold, on patients' daily lives.
  Each item is rated on a Likert-type scale from 0 to 7.
  0 = no symptoms / not at all
  7 = very severe / very much

OTHER OUTCOMES:
Incidence and severity of Adverse Events | 16 weeks
  Incidence and severity of all Adverse Events during the study (treatment and follow up period) related or not with the study product

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Taverniti, Microbes & Health R&D Leader, Study Director — Centro Sperimentale del Latte S.r.l.
Locations (1):
- Universidad Católica San Antonio de Murcia (UCAM), Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No